CLINICAL TRIAL: NCT00398814
Title: An Open-Label Phase I Study of the Safety of Perifosine in Combination With Sorafenib for Patients With Advanced Cancers
Brief Title: Phase I Study of Perifosine + Sorafenib for Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 124
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2011-11

CONDITIONS: Renal Cancer; Tumors
Keywords: Perifosine; Sorafenib; Renal cancer; Hepatocellular cancer; other advanced solid tumors
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms; Liver Neoplasms | interventions — perifosine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perifosine + Sorafenib (Experimental)
  Interventions: Drug: Perifosine; Drug: Sorafenib

INTERVENTIONS:
Drug: Perifosine — For the purposes of this study, one cycle of therapy will be defined as 4 weeks. Patients will take perifosine one to three times a day and will also receive sorafenib one to two times a day.
Drug: Sorafenib — For the purposes of this study, one cycle of therapy will be defined as 4 weeks. Patients will take perifosine one to three times a day and will also receive sorafenib one to two times a day.

SUMMARY:
This study is a Phase I trial in two parts. In part 1, a MTD to the combination of perifosine and sorafenib will be determined. In part 2, with the MTD as a starting point, a group of patients will be accrued with the goal of ensuring that they will be able to tolerate at least three courses of therapy, which would make them evaluable for response in a Phase II study.

DETAILED DESCRIPTION:
This study is a Phase I trial in two parts. In part 1, an MTD to the combination of perifosine and sorafenib will be determined. The experience with perifosine and other biologic agents has been that doses determined in Phase I studies are not as well tolerated in larger groups of patients when response is an endpoint. Thus in part 2, with the MTD as a starting point, a group of patients will be accrued with the goal of ensuring that they will be able to tolerate at least three courses of therapy, which would make them evaluable for response in a Phase II study. The effects of the combination of perifosine and sorafenib will be evaluated for response rate and time to progression. The pharmacokinetics of the combination of the study drugs will be measured.

For the purposes of this study, one cycle of therapy will be defined as 4 weeks. Patients will take perifosine one to three times a day and will also receive sorafenib one to two times a day. Patients may need anti-emetics and/or anti-diarrheals.

* Patients who experience toxicity may continue on treatment with doses delayed or reduced.
* All patients should continue therapy unless disease progression is documented on two occasions four weeks apart

All patients should be evaluated at each visit for adverse events. Patients will keep a diary documenting compliance with study drug, toxicities and any symptoms of hand/foot syndrome including numbness, tingling, redness or presence of sores, and any symptoms of hypertension. Patients will be evaluated for progression or response at 12-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically confirmed diagnosis of renal or hepatocellular tumor are eligible for this protocol. Patients with other solid tumor types must have their cases reviewed by the medical monitor.
* The physician must believe that the patient's course and the growth rate of the tumor are such that the patient would feel comfortable continuing treatment for 12 weeks even if there is a transient period of modest tumor growth during the first weeks following the initiation of perifosine and sorafenib treatment.
* Patients must have a life expectancy of more than 6 months.
* Patients may have received prior sorafenib or sunitinib malate.
* Patients may have measurable or evaluable disease.
* Patients should have a performance status of 0 to 1 according to the ECOG criteria.
* Patients must have adequate organ and marrow function, unless in the opinion of the treating investigator, the abnormality is related to tumor and the medical monitor agrees the abnormality is unlikely to affect the safety of perifosine use.
* Patients must have recovered from acute toxicity related to prior therapy including surgery or radiotherapy, excluding alopecia.
* Patients with breast cancer or prostate cancer who discontinue endocrine therapy prior to entry onto this study must wait for a minimum of 1 month and then be reassessed for a withdrawal response prior to starting perifosine. However, it is not a requirement that endocrine therapies be discontinued.
* Patients must be able to ingest oral medications or to obtain them through a gastrostomy tube.
* Patients must be at least 18 years of age.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Rapidly progressing disease, as defined by progression within 12 weeks of initiation of the previous regimen (see Section 8.2.8 below)
* Patients who have had more than three prior systemic therapies, including biologics, are excluded unless prior approval is obtained from the medical monitor.
* Patients receiving any other investigational agents or devices
* Patients initiating treatment for their cancer within the last two months who will be continued concomitantly with perifosine
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), or New York Heart Association class II-IV congestive heart failure
* Female patients who are pregnant or lactating are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Toxicity | Monthly

SECONDARY OUTCOMES:
Response or progression | 6 months

REFERENCES:
- [Result] Preliminary results / Journal of Clinical Oncology, 2008 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 26, No 15S (May 20 Supplement), 2008: 16024